CLINICAL TRIAL: NCT02678507
Title: A Quantitative Study to Assess the Construct Validity of the Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)
Brief Title: A Quantitative Study to Assess the Construct Validity of the Prescription Opioid Misuse and Abuse Questionnaire
Acronym: POMAQ
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: Evidera (Industry)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-4; 3033-4 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with chronic pain on opioids
  Interventions: Other: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)

INTERVENTIONS:
Other: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)

SUMMARY:
The purposes of this study are to evaluate the validity and reproducibility of the POMAQ to identify opioid abuse and misuse behaviors among participants who have chronic pain which requires long-term opioid use.

DETAILED DESCRIPTION:
The Food and Drug Administration (FDA) has requested, as part of a Post-marketing requirement (PMR) for new drug application (NDA) holders of extended release/long-acting (ER/LA) opioids, to conduct a study to develop and validate a measure of the opioid-related adverse events misuse and abuse among patients with chronic pain prescribed long-term opioid therapy. This measure will be used to assess misuse and abuse in PMR Study 2065-1A and PMR Study 2065-4B.

To date, no tool currently exists to address the needs of the PMR except for the Self-Report Misuse, Abuse and Diversion of Prescription (Rx) Opioids questionnaire (SR-MAD) which has undergone several rounds of content validation but requires further validation. The SR-MAD has been substantially modified to meet the needs of PMR Studies 2065-1A and 2065-4B and has been renamed the Prescription Opioid Misuse and Abuse Questionnaire (POMAQ). The POMAQ will undergo content validation via qualitative interviews (Protocol 2065-2A [Qualitative]) prior to use in this validation study (Protocol 2065-2A [Quantitative]).

This quantitative study will seek to further develop and validate the POMAQ following the general tenants according to the Food and Drug Administration (FDA) Guidance for Industry, Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims (FDA 2009) which emphasizes the importance of conducting sound psychometric evaluation of patient-reported instruments through quantitative research methods. However, it should be noted that the POMAQ is not a typical PRO measure capturing a specific latent construct and the specified analytic approach to the POMAQ reflects this difference in theoretical frameworks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Diagnosed chronic pain (≥ 3 months) condition which requires long-term treatment with opioids;
3. Willingness to provide written informed consent; and
4. Able to participate in and complete an Internet-based survey and a telephone interview in English.

Exclusion Criteria:

1. Cognitive or other impairment based on the Principal Investigator's judgment that would interfere with the ability of a participant to complete the validation study
2. Terminal illness with life expectancy <6 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients within the Department of Defense (DoD)/TriCare health system with chronic (>3 months) pain treated with opioids.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Identification Validity of the POMAQ in misuse and abuse of prescription opioid behaviors | Single Survey, with re-test in 20% of population 7-10 days after initial completion

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Barsdorf, Ph.D., Study Chair — Pfizer